CLINICAL TRIAL: NCT06347848
Title: The Effect of Psychoeducation Focused on Reducing Internalized Stigma in Individuals Diagnosed With Schizophrenia on Treatment Adherence and Internalized Stigma
Brief Title: The Effect of Psychoeducation Focused on Reducing Internalized Stigma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kadriye Atar, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulUCKA
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia; Treatment Adherence; Stigma, Social
Keywords: Schizophrenia; Treatment Adherence; Internalized Stigma; Psychoeducation
MeSH Terms: conditions — Schizophrenia; Treatment Adherence and Compliance; Social Stigma

STUDY DESIGN:
Intervention Model Description: Two parallel groups randomized control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Psyhcoeducation Group (Experimental) Psychoeducation focused on reducing internalized stigma will be applied to the experimental group.
  Interventions: Other: Psychoeducation Focused on Reducing Internalized Stigma
- No Intervention (No Intervention): Controls (Control Group) No intervention will be applied to the control group.

INTERVENTIONS:
Other: Psychoeducation Focused on Reducing Internalized Stigma — Participants will be randomized and divided into experimental and control groups. Initial measurements will be collected through a face-to-face meeting. While the control group will continue to receive routine Community Mental Health Center service, the experimental group will receive a psychoeducation program focused on reducing internalized stigma in addition to the routine Community Mental Health Center service. After the program is completed, final measurements of the experimental and control groups will be collected.
  The program is planned to consist of 7 sessions, once a week, and approximately 60-90 minutes are expected to be allocated for each session. Sessions will be divided into two sessions: a 30-40 minute session and a 15 minute break.
  Arms: Experimental

SUMMARY:
In the fight against stigma, the focus should be on the education of individuals diagnosed with mental illness. Psychoeducation has an important place in the treatment and rehabilitation of mental health problems. Psychoeducation is necessary for early recognition of signs and symptoms of diseases, ensuring compliance with treatment, improving coping skills, as well as combating stigma, preventing internalized stigma, and counteracting social stigma. If individuals with mental disorders have adequate knowledge about the causes of stigma, they may be less prone to internalized stigma.

DETAILED DESCRIPTION:
The group most exposed to stigma among mental illnesses is individuals diagnosed with schizophrenia. These individuals avoid treatment due to fear of stigma, which creates a significant obstacle to ensuring their well-being. Internalization of stigma causes feelings of loneliness, anger, helplessness, deterioration in quality of life, and decrease in self-esteem, while at the same time creating a significant barrier to treatment compliance. Compliance problems with treatment: It causes impairments in functionality, relapses and exacerbations, repeated hospitalizations, adverse effects on quality of life and increased mortality rates. The fact that many patients who receive only medical treatment in the treatment of schizophrenia develop negative attitudes towards drug use due to drug side effects and recurrence of disease symptoms reveals that psychosocial approaches should also be given importance in addition to medical treatment. As a result, it is thought that internalized stigma is a significant obstacle to treatment compliance and practices implemented to reduce internalized stigma are effective in increasing treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Diagnosed with schizophrenia according to DSM-V TR diagnostic criteria,
* Over 18 years old,
* Being in remission for 2 months,
* At least primary school graduate,
* Residing in Edirne city center and its districts,
* Individuals without hearing or understanding problems.

Exclusion Criteria:

* Not meeting the inclusion criteria,
* Having a diagnosis of dementia or other organic mental disorder as an additional diagnosis,
* Individuals with a history of substance abuse (other than nicotine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Internalized Stigma of Mental Illness Scale | 4 Month
  It is a self-report scale consisting of 29 items and assessing internal stigma. The scale includes: 1. Alienation (6 items), 2. Endorsement of Stereotypes (7 items), 3. Perceived Discrimination (5 items), 4. Social Withdrawal (6 items) and 5. Resistance to Stigma (5 items). It has five subscales. The items in the scale are on a four-point Likert-type scale as "I strongly disagree" (1 point), "I disagree" (2 points), "I agree" (3 points), "I strongly agree" (4 points). is answered. Items of the "Resistance to stigma" subscale are scored reversely.
  The total score obtained by summing the scores of the five subscales varies between 29 and 116 points. Higher scores from the scale mean that the person's internalized stigma is more severe in a negative way. While the internal consistency coefficient obtained for the entire scale was found to be 0.93, the split-half reliability of the scale was determined as 0.89.
Medication Adherence Reporting Scale | 4 Month
  It is a 5-point Likert type scale consisting of 5 questions. The scale is used to evaluate medication compliance in many diseases such as blood pressure, diabetes, rheumatoid arthritis, inflammatory bowel disease, hyperlipidemia, chronic pain, and bipolar mood disorder. The total test score is obtained by adding the scores obtained from the items. Scores from the scale vary between 5 and 25. An increase in the scores obtained indicates compatibility, and a decrease in the scores indicates non-compliance. It was found that the scale was evaluated with a single factor structure and had good levels of criterion and discriminant validity and reliability (Cronbach Alpha = 0.85).

CONTACTS AND LOCATIONS:
Overall Officials: Ozge SUKUT, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No